CLINICAL TRIAL: NCT03521726
Title: Visiting Staff, Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan
Brief Title: Intraluminal Amoxicillin Powder Monotherapy for Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tai-cherng Liou, MD, Principle investigator, Mackay Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17MMHIS096
Record Dates: First submitted 2018-04-22; First posted 2018-05-11 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Rabeprazole; Amoxicillin; Helicobacter Pylori
MeSH Terms: interventions — Amoxicillin; Rabeprazole

STUDY DESIGN:
Intervention Model Description: 20 participants receive intraluminal eradication of H. pylori. Patients fail to achieve intraluminal eradication of H. pylori will be assigned to the oral antibiotic rescue therapies with High-dose PPI-amoxicillin dual therapy (rabeprazole 20 mg and amoxicillin 750 mg 4 times/day) for 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraluminal Amoxicillin eradication (Other): 20 Patients receive intraluminal Amoxicillin eradication of H. pylori.
  Interventions: Drug: Amoxicillin
- Rabeprazole, Amoxicillin dual therapy (Other): Patients fail to achieve intraluminal eradication of H. pylori will be assigned to the oral antibiotic rescue therapies with high dose dual therapy (Rabeprazole and Amoxicillin) for 14 days.
  Interventions: Drug: Rabeprazole, Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Twenty patients receive Intraluminal Amoxicillin eradication for H. pylori.
  Other Names: Supercillin
  Arms: Intraluminal Amoxicillin eradication
Drug: Rabeprazole, Amoxicillin — Patients fail to achieve intraluminal eradication of H. pylori will be assigned to the oral antibiotic rescue therapies with high dose dual therapy (Rabeprazole, Amoxicillin) for 14 days.
  Other Names: Pariet, Supercillin
  Arms: Rabeprazole, Amoxicillin dual therapy

SUMMARY:
Helicobacter pylori (H. pylori) is the most common chronic bacterial infection in humans.

The prevalence of H. pylori is about 30~50% in the Western adult population. It is estimated that about 50% of people are infected with this bacterium in Taiwan. Many studies have shown that H. pylori is an important causal factor of chronic gastritis, peptic ulcer disease, gastric cancer and gastric lymphoma. The World Health Organization classified H. pylori as a Group 1 carcinogen in 1994. Endoscopic examination is indicated to confirm the above diagnosis for patient with H. pylori infection. Eradication of H. pylori infection reduces the risk of gastric cancer and recurrence of peptic ulcer disease. However, the eradication rate of clarithromycin-based triple therapy has been declining in recent years, probably related to the increasing resistant rate to clarithromycin. Several strategies have been proposed to overcome the declining eradication rate, including (1) extending the treatment duration of triple therapy to 14 days; (2) the use of bismuth quadruple therapy which contains bismuth, a proton pump inhibitor, and two antibiotics (usually metronidazole and tetracycline); (3) non-bismuth quadruple therapy (concomitant therapy) which contains a proton pump inhibitor and three antibiotics (usually amoxicillin, metronidazole, and clarithromycin); (4) sequential therapy which contains a proton pump inhibitor (PPI) plus amoxicillin for five days, followed by a PPI plus clarithromycin and tinidazole for another five days. The investigators aim to evaluate the efficacy of Amoxicillin powder in the Intraluminal therapy for Helicobacter pylori infection while an endoscopic examination is performed.

DETAILED DESCRIPTION:
During the endoscopic examination, patient is sedated with intravenous Dormicum 5mg (5mg/1ml/amp), the vital signs will be closely monitored by physiological monitor (PHILIPS SureSigns VM6). The treatment will be terminated immediately if unstable vital sign detected or if patient asks for termination. Patients will receive test for UFT300 to evaluate H. pylori colonization in the gastric cardia. With endoscope apparatus, the gastric mucous is irrigated with acetylcysteine solution and the pH value of gastric juice will be measured with the pH test strips before irrigation and after irrigation. The investigators dispense medicaments containing Amoxicillin powder in the capsule (3 gm) on the surface of gastric mucosa and duodenal mucosa of duodenal bulb as evenly as possible. After the intraluminal therapy, patients will rest for 30 to 60 minutes and go home if the effect of sedation subsided. Patients can take meal if no abdominal discomfort. C13-Urea breath test (UBT) will be used to assess the existence of H. pylori 6 weeks after the intraluminal therapy. Patients fail to achieve intraluminal eradication of H. pylori will be assigned to the oral antibiotic rescue therapies with High-dose PPI-amoxicillin dual therapy (rabeprazole 20 mg and amoxicillin 750 mg 4 times/day) for 14 days. C13-UBT will be used to assess the existence of H. pylori 6 weeks after the rescue therapy. Overall eradication rates after the first line intraluminal therapy and the oral antibiotics rescue therapies will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged greater than 20 years and less than 75 years
2. Patients have H. pylori infection without prior eradication therapy
3. Patients are willing to receive the intraluminal therapy. The written informed consents will be obtained from all patients prior to enrollment.

Exclusion Criteria:

1. Children and teenagers aged less than 20 years, and adult greater than 75 years
2. Contraindication for endoscopic examination or food retention in the gastric lumen.
3. History of gastrectomy; Gastroduodenal stenosis、deformity or obstruction; Gastroduodenal malignancy, including adenocarcinoma and lymphoma
4. Contraindication to treatment drugs: previous allergic reaction to amoxicillin, Proton pump inhibitors (lansoprazole, rabeprazole), Acetylcystein and Sucralfate; pregnant or lactating women
5. Severe concurrent acute or chronic illness: renal failure, cirrhosis of liver, incurable malignant disease
6. Patients who cannot give informed consent by himself or herself.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Eradication rate in the intraluminal therapy | 6 weeks after finishing therapy
  Eradication rate in the intraluminal therapy C13-UBT will be used to assess the existence of H. pylori 6 weeks after the intraluminal therapy.

SECONDARY OUTCOMES:
Overall eradication rates | 3-6 months after finishing intraluminal therapy
  Overall eradication rates after the first line intraluminal therapy and the oral antibiotics rescue therapies.

OTHER OUTCOMES:
Incidence of adverse effects in the intraluminal therapy. | within 7 days after finishing the intraluminal therapy
  Incidence of adverse effects were evaluated for Participants who had or had not finished the intraluminal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tai-cherng Liou, MD, Principal Investigator — Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital
Locations (1):
- Division of Gastroenterology and Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No